CLINICAL TRIAL: NCT06591208
Title: Study the Effect of Pulsed Dye Laser Versus Carboxytherapy in the Treatment of Striae Rubra
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aya Mohamed Fahim, principle investigator, Cairo University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: effect PDL vs carboxy on stria
Record Dates: First submitted 2024-09-09; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Striae Distensae
MeSH Terms: conditions — Striae Distensae | interventions — Lasers, Dye

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- single group 20 patients subjected PDL on one randomized side and carboxytherapy on the other side (Other)
  Interventions: Device: pulsed dye laser; Device: Carboxytherapy

INTERVENTIONS:
Device: pulsed dye laser — PDL (Cynosure - Chelmsford, MA-USA) wavelength 585 nm at a fluence 2.5-5 J/cm2, pulse duration of 0.5 ms and spot size 7 -10 mm
Device: Carboxytherapy — carboxytherapy (Carbo - Programmable automatic carbon dioxide therapy apparatus, MA-USA) that was automatically calibrated to adjust the flow rate, through regulation of infusion pressure and the dosage of CO2 in ml. the infusion velocity consequently was adjusted to a flow rate of 1 cc/. The injection performed slowly, subcutaneously, by tilting the needle at 15 degree using a sterile disposable insulin needle, with the depth adjusted at 2 mm. the gas volume per injection spot is 2ml with 1.5 cm spacing between each injection point. End point was skin distension with the gas giving the characteristic "popcorn appearance".

SUMMARY:
This clinical intrapatient randomized trial will be conducted on 20 patients of both genders complaining from bilateral symmetrical striae rubra. They will be recruited from Outpatient Clinic of Dermatology Department of Cairo University Hospitals. All included patients will be subjected to:

1. Informed written consent will be taken from every patient including the study.
2. Detailed history including onset, course, duration of the disease and occupation, predisposing factors, associated diseases and previous treatments.
3. Outcome will be done at baseline, after the last session and 2 months after the last session:

   * Photographing documentation: two photographs (in appropriate views) will be taken on two occasions; before each session (Baseline), and 2 months after the last treatment session.
   * Modified Vancouver Scar Scale The modified Vancouver Scar Scale (mVSS 1) evaluates four indicators: vascularity, pigmentation, pliability and height It has a score ranging from 0-13 The modified Vancouver Scar Scale (mVSS 2) evaluates three indicators: vascularity, pliability and height It has a score ranging from 0-10
   * Dermaspectrometer Dermaspectrometer will be measure erythema index at baseline, after the last session and 2 months after the last session.
   * Histopathological Assessment Skin biopsies using 4 mm punch biopsies will be obtained from SR before treatment (baseline) and 2 months after the last treatment sessions. The post-treatment biopsy will be taken from the vicinity of the baseline biopsy. Tissues will be fixed in 10% buffered formalin, will be embedded in paraffin and will be sectioned into 5 µm-thick sections. Specimens will be stained with hematoxylin and eosin (H & E) and/or Orcein (for demonstration of elastic fibers). Histological evaluations will be carried out under a light microscopy.

Pathologic assessment for the stria will be evaluated each of the epidermis, dermis, collagen fibers and elastic fibers. Degree of improvement will be assessed by examining the following criteria.

A.Epidermis: Epidermal thickness and presence of rete ridges B.Dermis: Papillary dermal edema, dermal vascularity, and presence of skin appendages.

C.Collagen fibers will be assessed for its thickness, commenting on whether it's fibrillar, fine thickness, normal thickness or sclerotic, besides the presence of perpendicular blood vessels towards the epidermis.

D.Elastic fibers: will be evaluated it through Orcein stain for its presence or absence, its thickness if present; fragmented or fibrillar.

* Blinded investigator evaluation

Two independent blinded investigators will be assessed clinical improvement. Assessment of the standardized photographs using the following score:

-1 = worse, 0 = no change,

1. = weak (1-24% improvement in striae),
2. = moderate (25-49% improvement in striae),
3. = good (50-74%improvement in striae)
4. = excellent (75-100% improvement in striae)

   * Patients' satisfaction

The patients' self-satisfaction for each modality of treatment (regarded improvement and side effects of each modality) measured on a five-point scale:

0 → not satisfied,

1. → moderately satisfied,
2. → satisfied, Treatment Protocol Twenty patients will be subjected to Pulsed Dye Laser (PDL) on one randomized side of their bodies and carboxytherapy on the other side for four sessions with four weeks' interval between sessions. Randomization will be done through picking red (PDL) yellow (carboxytherapy) cards.

After taking photographs, patients will be locally anesthetized by topical lidocaine under occlusion for 1 h on the side of carboxytherapy. The cream will be wiped off with a wet gauze when the session started. Protective eye wear will be provided to the patient, treating doctor and all the personnel assisting the procedure.

One randomized side of the affected area will be assigned to PDL (Cynosure - Chelmsford, MA-USA) with wavelength 585 nm at a fluence 2.5-5 J/cm2, pulse duration of 0.5 ms and spot size 7 -10 mm according to the width of the striae.

The other side will be assigned to carboxytherapy (Carbo - Programmable automatic carbon dioxide therapy apparatus, MA-USA) that will be automatically calibrated to adjust the flow rate, through regulation of infusion pressure and the dosage of CO2 in ml. the infusion velocity consequently will be adjusted to a flow rate of 1 cc/sec. The injection will be performed slowly, subcutaneously, by tilting the needle at 15 degree using a sterile disposable insulin needle, with the depth adjusted at 2 mm. the gas volume per injection spot is 2ml with 1.5 cm spacing between each injection point.

Each patient will be received 4 sessions with 4 weeks' intervals.

ELIGIBILITY:
Inclusion Criteria:

* 1. Both genders are included. 2. Patients above 18 years old. 3. Patients have bilateral symmetrical striae rubra lesions.

Exclusion Criteria:

1. Pregnancy
2. Scarring and keloid tendencies.
3. Active skin infection, active infection of herpes simplex virus.
4. Patient on Prior steroid therapy
5. Patient have History of Cushing syndrome
6. Patients with concomitant disease during the study (e.g., hepatic, renal, cardiac, autoimmune diseases, diabetes mellitus, and/or bleeding disorders).

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-09-11 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Patient Evaluation(mVSS Score, blinded investigators evaluation) | 6 months
  * Modified Vancouver Scar Scale The modified Vancouver Scar Scale (mVSS 1) evaluates four indicators: vascularity, pigmentation, pliability and height It has a score ranging from 0-13 The modified Vancouver Scar Scale (mVSS 2) evaluates three indicators: vascularity, pliability and height It has a score ranging from 0-10 Assessment for all patients will be at baseline after last session, and 2 months after last session.
  * Blinded investigator evaluation
  Two independent blinded investigators will be assessed clinical improvement. Assessment of the standardized photographs using the following score:
  -1 = worse, 0 = no change,
  1. = weak (1-24% improvement in striae),
  2. = moderate (25-49% improvement in striae),
  3. = good (50-74%improvement in striae)
  4. = excellent (75-100% improvement in striae

CONTACTS AND LOCATIONS:
Overall Officials: Rana Fathy Helal, assistant professor, Principal Investigator — Cairo University; Aya mohamed fahim, assistant professor, Principal Investigator — Cairo University

IPD SHARING:
Plan to Share IPD: Yes
results and discussion can be shared
Time Frame: after finishing the paper and and will be always available
Access Criteria: through the pubmed

REFERENCES:
- [Background] Hodeib AA, Hassan GFR, Ragab MNM, Hasby EA. Clinical and immunohistochemical comparative study of the efficacy of carboxytherapy vs platelet-rich plasma in treatment of stretch marks. J Cosmet Dermatol. 2018 Dec;17(6):1008-1015. doi: 10.1111/jocd.12481. Epub 2018 Jan 7. PMID 29316152
- [Background] Shokeir H, El Bedewi A, Sayed S, El Khalafawy G. Efficacy of pulsed dye laser versus intense pulsed light in the treatment of striae distensae. Dermatol Surg. 2014 Jun;40(6):632-40. doi: 10.1111/dsu.0000000000000007. PMID 24852467